CLINICAL TRIAL: NCT06794346
Title: Effects of Vaginal or Transdermal Testosterone on Sexual Response and Climacteric Symptoms in Postmenopausal Women
Brief Title: Sexual Effects of Transdermal or Vaginal Testosterone
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Jose Maria Soares Junior, Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2907493
Record Dates: First submitted 2022-03-18; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-04

CONDITIONS: Female Sexual Dysfunction; Postmenopausal Symptoms; Testosterone Deficiency; Testosterone Adverse Reaction
Keywords: Sexual effects of transdermal or vaginal testosterone; low sexual desire; postmenopause; transdermal testosterone; vaginal testosterone

STUDY DESIGN:
Intervention Model Description: This is a phase 2, randomized, double-blind, parallel-group clinical trial with a 24-week follow-up of patients using testosterone 300 mcg (transdermal or vaginal cream) versus placebo.
  The patients will be distributed as follows:
  Group A : will receive transdermal testosterone (300 mcg) and vaginal placebo for 24 weeks Group B : will receive transdermal placebo and vaginal testosterone (300 mcg) for 24 weeks Group C: will receive transdermal and vaginal placebo for 24 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients are randomized into 3 different groups and given a number 1 to 132 to identify wich arm is she in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transdermal testosterone (Experimental): In this group women will receive vaginal placebo cream and transdermal testosterone cream (300mcg)
  Interventions: Drug: Transdermal testosterone
- Vaginal testosterone cream (Experimental): In this group women will receive vaginal testosterone cream (300 mcg) and transdermal placebo cream
  Interventions: Drug: Vaginal testosterone gel
- Placebo (Placebo Comparator): In this group women will receive vaginal placebo cream e transdermal placebo cream
  Interventions: Device: Placebo group

INTERVENTIONS:
Drug: Transdermal testosterone — women will receive 300mcg of transdermal testosterone in cream daily for six months
  Other Names: transdermal group
  Arms: Transdermal testosterone
Drug: Vaginal testosterone gel — women will receive 300mcg of vaginal gel testosterone daily for six months
  Other Names: vaginal group
  Arms: Vaginal testosterone cream
Device: Placebo group — women will receive both vaginal gel and transdermal cream placebo for six months
  Arms: Placebo

SUMMARY:
The aim of the study is to elucidate the role of testosterone treatment in postmenopausal women's sexual function and their therapeutic safety.

DETAILED DESCRIPTION:
-General To evaluate the therapeutic efficacy of testosterone treatment in sexual dysfunction in postmenopausal patients.

-Specifics

1. To evaluate the prevalence of different sexual dysfunctions in postmenopausal patients, classifying them according to Diagnostic and Statistical Manual of Mental Disorders 5th (2013):

   * Female sexual desire / arousal disorder;
   * Female orgasm disorder;
   * pelvic or genital pain / penetration disorder;
2. To evaluate the response on climacteric symptoms after testosterone replacement using the Kupperman Menopausal Index;

ELIGIBILITY:
Inclusion Criteria:

* Brazilian women with menopause time from 2 to 6 years;
* active sex life;
* absence of severe depression and anxiety, as evidenced by the Beck (depression specific) and Beck (anxiety specific) questionnaires;

Exclusion Criteria:

* disabling diseases;
* use of medicines that inhibit sexual desire;
* inability to answer the questionnaires;
* altered routine exams and comorbidities:

  * Severe hypertension with Blood Pressure measurement > 160 mmHg (maximum) or/and 90 mmHg (minimum) in two measurements
  * clinical or subclinical thyroid dysfunction: thyroid-stimulating hormone over 4
  * triglyceride dyslipidemia> 400
  * presence of occult blood in stool
  * hyperprolactinemia
  * fasting blood glucose> 100
  * presence of osteopenia or osteoporosis
  * BIRADS score greater than or equal to 3 on mammography
  * presence of endometrial echo> 4mm on transvaginal ultrasound
  * Presence of changes in oncotic colpocytology
* Diagnosis after psychological screening for moderate to severe anxiety / depression.

Ages: 38 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female self-identified gender are accepted for the study
Enrollment: 132 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in sexual disorders measured by FSFI (Female Sexual Function index) after 12 and 24 weeks of treatment | From enrollment to the end of treatment at 24 weeks
  We expect a 40% change for better in sexual complaints for the experimental group when compared with the placebo group.
  We will use the FSFI questionaire (Female sexual function index): a multidimensional self-Report instrument for the assessment of female sexual function (including desire/ libido, arousal, pain/discomfort, and orgasm) translated and validated to portuguese applied on time 0, 12 weeks and 24 weeks for each patient.
  Cite: Pacagnella RC, Martinez EZ, Vieira EM. Cad. Saúde Pública, Rio de Janeiro; 25 (11): 2333-2344. Nov 2009.

SECONDARY OUTCOMES:
Changes in hypoactive desire and arousal measured by FSFI ( Female Sexual Function Index) after 12 and 24 weeks of treatment | From enrollment to the end of treatment at 24 weeks
  We expect a 40% change for better in hypoactive desire and arousal complaints in the group that receive testosterone, either the transdermal or vaginal .
  We will use the FSFI (Female sexual function index) translated and validated to portuguese to access the desire/libido before, during and after intervention.
  Cite: Pacagnella RC, Martinez EZ, Vieira EM. Cad Saúde Pública, Rio de Janeiro; 25(11): 2333-2344, Nov 2009.
Change in orgasm measured by FSFI ( Female Sexual Function Index) after 12 and 24 weeks of treatment | From enrollment to the end of treatment at 24 weeks
  We expect a 40% change for better in orgasm complaints in the group that receive testosterone, either the transdermal or vaginal . We will use the FSFI (Female sexual function index) translated and validated to portuguese to access changes in orgasm before, during and after intervention. Cite: Pacagnella RC, Martinez EZ, Vieira EM. Cad Saúde Pública, Rio de Janeiro; 25(11): 2333-2344, Nov 2009
change in genitopelvic pain measured by FSFI ( Female Sexual Function Index) after 12 and 24 weeks of treatment | From enrollment to the end of treatment at 24 weeks
  We expect a 40% change for better in pain complaints in the group that receive testosterone, either the transdermal or vaginal . We will use the FSFI (Female sexual function index) translated and validated to portuguese to access changes in orgasm before, during and after intervention. Cite: Pacagnella RC, Martinez EZ, Vieira EM. Cad Saúde Pública, Rio de Janeiro; 25(11): 2333-2344, Nov 2009
Change in climateric symptoms measured by Blatt-Kupperman Menopausal Index questionaire after 12 and 24 weeks of treatment | From enrollment to the end of treatment at 24 weeks
  We expect a 50% change for better of climateric symptoms complaints in the group that receive testosterone, either transdermal or vaginal .
  We will use Blatt-Kupperman menopausal índex questionnaire before, during and after the intervention.
  cite:
  1. Kupperman et al, Menopausal Syndrome. JAMA, 171 (12): 1627-1637. Nov 1959.
  2. Alder E. The Blatt-Kupperman Menopausal Index: a critique. Maturitas, 29(1): 19-24. May 1998.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund C Baracat, Head, Study Chair — University of Sao Paulo General Hospital
Locations (1):
- Flavia Fairbanks, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The study is still in progress and we don´t have the preliminary data available.

REFERENCES:
- [Background] Abdo CH, Oliveira WM Jr, Moreira ED Jr, Fittipaldi JA. Prevalence of sexual dysfunctions and correlated conditions in a sample of Brazilian women--results of the Brazilian study on sexual behavior (BSSB). Int J Impot Res. 2004 Apr;16(2):160-6. doi: 10.1038/sj.ijir.3901198. PMID 14961047
- [Background] Alexander JL, Dennerstein L, Burger H, Graziottin A. Testosterone and libido in surgically and naturally menopausal women. Womens Health (Lond). 2006 May;2(3):459-77. doi: 10.2217/17455057.2.3.459. PMID 19803917